CLINICAL TRIAL: NCT04129307
Title: Assessment of the Effects of Brain Training Tools in Combination With Physical Practice on the Acquisition of Different Motor Tasks: a Randomised Controlled Trial
Brief Title: Brain Training Tools With Physical Practice on Motor Learning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: uammadrid2
Record Dates: First submitted 2019-10-10; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Motor Learning
Keywords: Motor imagery; Action observation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor Imagery (Experimental)
  Interventions: Behavioral: Motor imagery
- Double time Motor imagery (Experimental)
  Interventions: Behavioral: Double time motor imagery
- Action observation (Active Comparator)
  Interventions: Behavioral: Action observation

INTERVENTIONS:
Behavioral: Motor imagery — This group will perform motor imagery training in combination with physical practice on motor learning of different motor tasks.
  Arms: Motor Imagery
Behavioral: Double time motor imagery — This group will perform motor imagery training by doubling the intervention time to the motor imagery group in combination with physical practice on motor learning of various motor tasks.
  Arms: Double time Motor imagery
Behavioral: Action observation — This group will perform action observation training in combination with physical practice on motor learning of various motor tasks.
  Arms: Action observation

SUMMARY:
This study evaluates the influence of motor imagery and action observation in combination with physical practice on motor learning

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic subjects
* men and women between 18 and 65 years of age
* participants with no systemic, neurological, cognitive or psychological disease.

Exclusion Criteria:

* underage participants
* presence of systemic pathology, pain and/or weakness that prevents the protocol
* participants who have undergone an operation in the spine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Hit ratio in a manual skill test | Change from hit ratio in a manual skill at 1 week
  This main variable will be composed by the learning of a sequence of digital movements.
Free basketball shots | Change from hit ratio in free throws at 1 week
  The percentage of successful basketball shots in different positions will be counted.
Standing jump | Change from distance at 1 week
  Subjects shall place their feet shoulder width apart and their toes in a line on the floor. The subjects will then make a horizontal leap forward, where they are allowed to swing their arms along a tape measure attached to the floor.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No